CLINICAL TRIAL: NCT02977806
Title: The Evaluation of Iron Metabolism Using a Novel Isotope Dilution Method in Malawian Children, Who Have Previously Participated in a Stable Isotope Study
Brief Title: Iron Long-Term Labelling Study Malawi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Michael B. Zimmermann (Other)
Responsible Party: Sponsor-Investigator, Prof. Michael B. Zimmermann, Professor, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: Fe_LTL_Ma
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Iron Absorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Conventional indirect indicators of iron status, using serum and red blood cell biomarkers, are confounded by inflammation from common infections in sub-Saharan Africa, a region with a high prevalence of iron deficiency, making the assessment of iron balance and efficiency of iron intervention difficult. A new method allowing accurate measurement of long-term oral iron absorption and allowing the estimation of iron requirements is highly needed. Such a novel method to quantify iron absorption and requirements using isotope dilution measurements in children should be validated in the present prospective observational study by following-up a group of 49 children given a stable iron isotope in an earlier trial. We will request seven blood samples within 2 years (sampling every four months) from the participants which will allow us to measure isotopic dilution for estimating total oral iron absorption over these 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in the original absorption study and the two follow-up samplings
* Signed written informed consent from the guardian to participate in the study

Exclusion Criteria:

* Long-term medication
* Any severe metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the guardian's statement or med-ical examination (health booklet))
* Blood losses (surgery, accident) or blood transfusion during the past 4 months before study start.
* Residence too far away (> 2 hours by motorbike) from study location (Zomba)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Malawian children who ingested stable iron isotopes in the frame of a former iron absorption study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
iron isotope composition in blood | 2 years
  the iron isotope ratio (tracer/tracee ratio) in blood should be analyzed with ICPMS every 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof., Principal Investigator — Human Nutrition Laboratory, ETH Zürich
Locations (1):
- College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No